CLINICAL TRIAL: NCT02057276
Title: Motor Control Enhancement Through Repetitive Transcranial Magnetic Stimulation Plus Rehabilitation in Hemiparetic Cerebral Palsy and Stroke
Brief Title: Repetitive TMS and Occupational Therapy in Children and Young Adults With Chronic Hemiparesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to low recruitment.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIN001 - rTMS/hemiparesis; 2012-1533 (Other: Cincinnati Children's Hospital Medical Center)
Record Dates: First submitted 2013-06-05; First posted 2014-02-07 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Pediatric Stroke; Cerebral Palsy; Chronic Hemiparesis
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Magnetic Stimulation; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS (Active Comparator): Participants will receive daily active rTMS with occupational therapy immediately following rTMS for 10 consecutive weekdays.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Other: Occupational Therapy
- Sham rTMS (Sham Comparator): Participants will receive daily sham rTMS with occupational therapy immediately following rTMS for 10 consecutive weekdays.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation; Other: Occupational Therapy

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — We will use a specific rTMS paradigm called Continuous Theta Burst Stimulation (cTBS) for this study.
  Arms: Active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation
  Arms: Sham rTMS
Other: Occupational Therapy

SUMMARY:
The purpose of this study is to determine whether Repetitive Transcranial Magnetic Stimulation (rTMS) can augment occupational therapy in improving motor function in children (10 years of age or older) and young adults (< 21 years of age) with chronic hemiparesis from either stroke or cerebral palsy.

DETAILED DESCRIPTION:
RTMS is a noninvasive technology that can induce changes in brain function that may lead to functional improvement in people with hemiparesis. This is a randomized, double-blinded, sham-controlled rTMS study in conjunction with intensive daily occupational therapy (OT) for 2 weeks to improve motor function in hemiparetic patients. Participants will be followed for at least 12 weeks after rTMS to detect any clinical change. The sham group participants will be offered an open-label active rTMS treatment plus OT after the 12 week assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 years; < 21 years
* Hemiparesis
* Manual Ability Classification System (MACS) level I through IV
* Provision of written informed consent by the patient and/or guardian, including understanding that insurance may be billed for the occupational therapy
* Written assent form signed by participants younger than 18 years of age

Exclusion Criteria:

* Underlying degenerative or metabolic disorder or supervening medical illness
* Severe depression or other psychiatric disorder
* Any participant who is pregnant
* Any contraindication to TMS (i.e., intracranial metal implants, shunts, ports, pacemaker, baclofen pumps)
* Any changes or addition of neuropsychiatric medications within 1 month of starting the study or during course of the study (if applicable)
* Any botulinum toxin (Botox, Myobloc) or phenol injection within the last 3 months prior to the study or during the course of the study (if applicable)
* Any upper extremity surgery within the last 6 months prior to the study or scheduled during the course of the study (if applicable)

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve W Wu, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Groups:
- Active rTMS: Participants will receive daily active rTMS with occupational therapy immediately following rTMS for 10 consecutive weekdays.
  Repetitive Transcranial Magnetic Stimulation: We will use a specific rTMS paradigm called Continuous Theta Burst Stimulation (cTBS) for this study.
  Occupational Therapy
- Sham rTMS: Participants will receive daily sham rTMS with occupational therapy immediately following rTMS for 10 consecutive weekdays.
  Sham Repetitive Transcranial Magnetic Stimulation
  Occupational Therapy
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
  Female |  |  | 0
  Male |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the "Melbourne Assessment of Unilateral Upper Limb Function"
Time Frame: Change in the "Melbourne Assessment of Unilateral Upper Limb Function" between baseline and 3 days after rTMS/OT
Population: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Change in the "Melbourne Assessment of Unilateral Upper Limb Function"
Time Frame: Change in the "Melbourne Assessment of Unilateral Upper Limb Function" between baseline and 7 days after rTMS/OT
Population: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Change in the "Melbourne Assessment of Unilateral Upper Limb Function"
Time Frame: Change in the "Melbourne Assessment of Unilateral Upper Limb Function" between baseline and 12 weeks after rTMS/OT
Population: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: After signing consent forms, two separate participants did not proceed with the study. The study was then terminated.
Arm/Group | Active rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes